CLINICAL TRIAL: NCT02893865
Title: Evolution of Oxidative Stress in Coronary Patients With Moderate Sleep Apnea Syndrome After Treatment With Continuous Positive Airway Pressure
Acronym: CardioX SAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9542
Record Dates: First submitted 2016-08-04; First posted 2016-09-09 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2021-10

CONDITIONS: Sleep Apnea Syndrome; Coronary Artery Disease
Keywords: Apnea syndrome; Coronary artery disease; Oxidative stress; Continuous positive airway pressure; Endothelial dysfunction
MeSH Terms: conditions — Sleep Apnea Syndromes; Coronary Artery Disease | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Continuous positive airway pressure Patients will receive continuous positive airway pressure during three months
  Interventions: Device: Continuous positive airway pressure
- Sham Comparator (Sham Comparator): Sham-continuous positive airway pressure Patients will receive sham-continuous positive airway pressure during 3 months
  Interventions: Device: Sham-continuous positive airway pressure

INTERVENTIONS:
Device: Continuous positive airway pressure — Continuous positive airway pressure treatment during three months with adherence recording
  Arms: Experimental
Device: Sham-continuous positive airway pressure — Sham-continuous positive airway pressure during three months with adherence recording
  Arms: Sham Comparator

SUMMARY:
Published data indicate that obstructive sleep apnea syndrome (OSAS) worse the prognosis of coronary artery disease (CAD) and that oxidative stress can link this 2 diseases.

Investigators hypothesise that oxidative stress decrease after 3 months of continuous positive airway pressure (CPAP) in this specific population.

The results may have major implication in the comprehension of physiopathologic processes linking OSAS and CAD and in the treatment of OSAS in this specific population.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) is a common disorder characterized by recurrent upper airway collapse during sleep and has been associated with worsened prognosis in patients with coronary artery disease (CAD). Moderate OSAS can be defined by an apnea hypopnea index (AHI) between 15 and 30 events/hour.

Pathophysiologic processes are complex and it seems that oxidative stress play and important role. Studies showed that continuous positive airway pressure (CPAP) influence oxidative stress but the results are conflicting.

Moreover there are uncertainties whether diagnosing and treating OSAS can inﬂuence the pathophysiological and clinical outcomes in patients with CAD.

Therefore, we aim to test the effects of 3 months of CPAP on systemic redox balance evaluated by plasma GSH/GSSG ratio.

Patients with moderate OSAS will be randomized for the intervention.

Patients with AHI <15/h or >30/h will be included in an ancillary study (blood and urinary test, MIBG scintigraphy) to characterize the biological profile of coronary patients based on their AHI.

For a alpha threshold of 5% and a study power of 80%, the study should include 16 patients in each group. Taking in account a possible 20% of dropout the study will need to include 20 patients by randomized arm to demonstrate an effect.

ELIGIBILITY:
Inclusion Criteria:

* Apnea Hypopnea Index 15-30/h
* Stable Coronary artery disease
* Obligation of obtaining informed consent form

Exclusion Criteria:

* Heart failure with LVEF less than or equal to 45%
* Other Chronic disease: renal failure, COPD Index - central apneas than or equal to 50% of the total IAH
* treatment with CPAP or mandibular advancement device
* IMC> 40 kg / m²
* Nutritional supplementation in the 4 weeks preceding the study (antioxidants, vitamins ...).
* Treatment with allopurinol or N-acetylcysteine, in the 4 weeks preceding the study.
* PaCO2> 45 mmHg - Counter-indication to the use of PPC: bullous lung disease, pathological hypotension, bypass airway, pneumothorax, signs of sinus infections or inner ear
* Exclusion period on subject compared to another protocol or for which the maximum annual amount of compensation of € 4,500 has been reached.
* Participation of the subject to another study.
* Not affiliated with a social security scheme subject or not the beneficiary of such a regime.
* Pregnant or breastfeeding women, patient unable to give consent, protected adult, vulnerable
* Subject deprived of liberty by judicial or administrative decision
* HIV infection, hepatitis B or hepatitis C known

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
Percentage change of serum GSH/GSSG ratio | at the inclusion and the end (3 months) of the study
  Blood test

SECONDARY OUTCOMES:
Change, after 3 months, of the SOD (parameter of serum oxidative stress level) | at the inclusion and the end (3 months) of the study
Change, after 3 months, of the catalase (parameters of serum oxidative stress level) | at the inclusion and the end (3 months) of the study
Change, after 3 months, of the Vit C and E (parameters of serum oxidative stress level) | at the inclusion and the end (3 months) of the study
Change, after 3 months, of the isoprostanes (parameter of serum oxidative stress level) | at the inclusion and the end (3 months) of the study
Change, after 3 months, of the 8OHDG (other parameters of serum oxidative stress level) | at the inclusion and the end (3 months) of the study
  by blood test
Change, after 3 months, of the GPX (parameter of serum oxidative stress level) | at the inclusion and the end (3 months) of the study
Change, after 3 months, of the inflammation parameters: IL6, IL8, TNF α (blood test) | at the inclusion and the end (3 months) of the study
Change, after 3 months, of the urinary catecholamines by urine test | at the inclusion and the end (3 months) of the study
Change, after 3 months, of the MIBG scintigraphy | at the inclusion and the end (3 months) of the study
Change, after 3 months, of the endothelial function (endoPat) | at the inclusion and the end (3 months) of the study
Change, after 3 months, of the blood pressure | at the inclusion and the end (3 months) of the study
  24h ambulatory blood pressure monitoring
Change, after 3 months, of the quality of life by the SF 36 questionnaire | at the inclusion and the end (3 months) of the study
Change, after 3 months, of the quality of sleep by PSQI questionnaire | at the inclusion and the end (3 months) of the study
Change, after 3 months, of the sleepiness by the Epworth scale | at the inclusion and the end (3 months) of the study
Change, after 3 months, of the physical activity by the Voorips questionnaire | at the inclusion and the end (3 months) of the study

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No